CLINICAL TRIAL: NCT01461577
Title: A Multicenter, Open-label, Single-arm, 24 Week Phase IV Study Evaluating the Effectiveness and Safety of Treatment of Insulin Glargine in Type 2 Diabetes Mellitus Following Glucagon-like Peptide-1 (GLP-1) Failure
Brief Title: Effectiveness and Safety of Treatment of Insulin Glargine in Type 2 Diabetes Mellitus Following Glucagon-like Peptide-1 (GLP-1) Failure
Acronym: GAUDI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_05477; U1111-1118-8753 (Other: UTN)
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- insulin glargine (Experimental): Insulin glargine will be administered once a day, in the morning, at initial dose of 4 units/day. Titration of insulin dose will be performed referred with the median fasting plasma glucose value for the last 3 consecutive days according to the titration algorithm
  Interventions: Drug: INSULIN GLARGINE HOE 901

INTERVENTIONS:
Drug: INSULIN GLARGINE HOE 901 — Pharmaceutical form:solution Route of administration: subcutaneous

SUMMARY:
Primary Objective:

* To assess the efficacy of insulin glargine as measured by changes of HbA1c levels from baseline in type 2 diabetes mellitus (T2DM) patients following GLP-1 failure.

Secondary Objective:

* To determine the change in glycemic control, safety, and treatment satisfaction in insulin glargine use in patients following GLP-1 failure.

DETAILED DESCRIPTION:
1-2 weeks screening period, 24 weeks treatment period, 1 week follow-up period

ELIGIBILITY:
Inclusion criteria:

* Patients of aged ≥30 and ≤75 years with type 2 diabetes mellitus (T2DM)
* Hemoglobin A1c (glycosylated hemoglobin; HbA1c) levels measured at screening ≥7.5%
* Continuous treatment with stable doses of GLP-1 analogue for >3 months prior to enrollment (for patients also using oral anti-hyperglycemic drugs [OADs], continuous treatment with stable doses of OADs for >3 months prior to enrollment)

Exclusion criteria:

* Inpatient with T2DM
* Diabetes other than T2DM (e.g. secondary to pancreatic disorders, drug or chemical agent intake)
* Fasting plasma glucose (FPG) levels <130mg/dL
* Body mass index (BMI) >28 kg/m2
* Patients using thiazolidinediones in the last 3 months prior to enrollment
* Use of any treatment for weight loss in the last 3 months prior to enrollment
* Treatment with systemic corticosteroids within the 3 months prior to enrollment
* Patients using non-selective ß-blockers
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical trial protocol
* Most recent ophthalmologic examination >6 months prior to enrollment
* Diabetic retinopathy with surgical treatment (last photocoagulation or vitrectomy) in the 3 months before enrollment or which may require surgical treatment
* Proliferative diabetic retinopathy or any other unstable rapidly progressive retinopathy
* Impaired renal function defined as, but not limited to, serum creatinine ≥1.3 mg/dL [males] or ≥1.2 mg/dL [females] or presence of macroproteinuria (>1 g/day)
* Active liver disease including hepatic cirrhosis, hepatic failure, and hepatitis or alanine transaminase (ALT) or aspartate aminotransferase (AST) >2 times upper limit or total bilirubin >1.5 times upper limit of normal (except in case of Gilbert's syndrome) at enrollment
* Have any condition (including known substance or alcohol abuse or psychiatric disorder) that precludes the patient from following and completing the study protocol
* Any medical condition that may have an influence on HbA1c rate
* Currently undergoing therapy for malignancy which may affect the study evaluation
* Use of any investigational product and/or device within the 2 months prior to enrollment
* History of ketoacidosis or hyperosmolar hyperglycemic state during the previous 12 months prior to enrollment
* History of stroke, myocardial infarction, angina pectoris, coronary artery bypass graft or percutaneous transluminal coronary angioplasty within the previous 12 months prior to enrollment
* History of congestive heart failure
* History of hypoglycemia unawareness or unexplained hypoglycemia during the previous 12 months prior to enrollment
* Hemoglobinopathy or hemolytic anemia, transfusion of blood or plasma products within 3 months prior to enrollment
* Known hypersensitivity / intolerance to insulin glargine or any of its excipients
* History of pancreatitis
* Pregnant or breast-feeding women (women of childbearing potential must have a negative pregnancy test at study entry and a medically approved contraception method)
* Shift workers or those who regularly work a night-time shift

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Efficacy assessment of insulin glargine measured by changes of HbA1c levels from baseline | 24 weeks

SECONDARY OUTCOMES:
Responder rate (HbA1c levels <7%) without severe hypoglycemia | 24 weeks
Responder rate (HbA1c levels <6.5% and <7%) | 24 weeks
Changes of fasting plasma glucose (FPG) levels from baseline | 24 weeks
Changes of beta cell marker: C-peptide from baseline | 24 weeks
Changes of Lipid profile: Lipid profile from baseline | 24 weeks
Weight change from baseline | 24 weeks
Total insulin dose (per kg body weight) | 24 weeks
Evaluation of patient's treatment satisfaction | 24 weeks
Number of patients with hypoglycemia | up to 24 weeks
Number of patients with treatment-emergent adverse events | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Administrative office, Tokyo, Japan